CLINICAL TRIAL: NCT05532579
Title: Effectiveness of an Invasive Physical Therapy Protocol in Primary Care Patients With Low Back Pain and Lower Extremity Irradiation. Randomized Controlled Clinical Trial
Brief Title: Effectiveness of an Invasive Physical Therapy Protocol in Primary Care Patients With Low Back Pain. Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jacobo Rodríguez Sanz, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFC22LBP
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invasive Physiotherapy (Experimental)
  Interventions: Other: Invasive Physiotherapy Group
- Sham Group (Placebo Comparator)
  Interventions: Other: Sham Group

INTERVENTIONS:
Other: Invasive Physiotherapy Group — The study participants corresponding to the intervention group will receive the treatment proposed by their medical doctor. In addition, and as the main part of the intervention, they will receive an invasive physiotherapy protocol consisting of 3 sessions of ultrasound-guided percutaneous neuromodulation, with a time margin of one week between the first and second session and two weeks between the second and third session. The session will last approximately 15 minutes. Each treatment session will consist of the application of a symmetric biphasic current of 3Hz frequency, 250µsec pulse width, 10 impacts of 10 seconds duration with 10 seconds of rest between them. This application will be performed with acupuncture needles placed in an echoguided manner in the proximity of the dorsal root of the last 3 lumbar levels and in the proximity of the sciatic nerve at its exit from the piriformis muscle.
  Arms: Invasive Physiotherapy
Other: Sham Group — Study participants corresponding to the sham group will receive the treatment proposed by their medical doctor. In addition, they will receive the application of the simulated transcutaneous electrical stimulation technique, placing the patches on the same points where the needles are located, remaining in prone position for the necessary time after the technique is performed until 15 minutes have elapsed. This technique has been studied as a placebo technique for neuromodulation interventions.
  Arms: Sham Group

SUMMARY:
Low back pain or lumbar pain is the most frequent cause of incapacity for work in Spain, occupying first place among the most common pathologies diagnosed in this country, followed by cervical pain. Non-specific low back pain is the main cause of public spending on health care and labor concepts, with a prevalence of 80%. Furthermore, this pathology represents more than half (52.92%) of the diagnoses of chronic pain that is neither oncologic nor neuropathic. This situation generates high economic, health care and labor costs, representing an equivalent cost of between 1.7% and 2.1% of the Gross Domestic Product.

Low back pain is described as pain located between the lower limit of the ribs and the lower limit of the buttocks, the intensity of which varies according to posture and physical activity, and which is usually accompanied by painful limitation of movement. Approximately 40% of patients with low back pain present irradiation in the lower extremity. The chronification of low back pain can result in central sensitization, causing hypersensitivity to non-painful and painful stimuli even long after the onset of the acute episode of low back pain.

The approach to low back pain offers options such as the administration of drugs, prescription of physical exercise, pain education and modification of patients' habits. Minimally invasive techniques in the management of low back pain are arousing greater interest due to their great advantages. In the field of physical therapy, novel techniques have been developed in recent years, such as ultrasound-guided percutaneous musculoskeletal electrolysis and ultrasound-guided percutaneous neuromodulation, in which different types of electric current are applied through solid needles. Different mechanisms of action have been associated with these invasive techniques, such as a potential effect on the activation of descending pain inhibitory system pathways, the reduction of evoked motor potentials and an increase in intracortical inhibition, suggesting benefits in patients with central sensitization. The invasive techniques of electrolysis and neuromodulation have been applied in other studies at the nervous level, especially in the sciatic nerve at the piriformis and ischiotibial level, in the popliteal fossa and in the foot. It has given good results in lumbar pain. However, there is no study carried out in patients with low back pain and the presence of hernias or protrusions, nor is there any control of the evolution in the medium and long term.

The application of percutaneous neuromodulation has the capacity to modulate neuronal activity in the primary motor cortex, promoting transient and long-term neuroplastic effects. The modulation of this region is related to a decrease in pain due to the relationship with pain processing areas, such as the thalamus, cingulate cortex and periaqueductal gray matter. Electrical stimulation of the peripheral nervous system percutaneously activates a complex neural network that in turn involves a series of neurotransmitters and receptors, such mechanisms being able to promote segmental analgesia and extra-segmental analgesia. Some studies suggest that percutaneous neuromodulation therapy may have a possible beneficial effect in patients with central sensitization, producing improved conditioned pain modulation, reduced motor evoked potential and enhanced intracortical inhibition.

To the authors' knowledge, there are no studies that prove the effectiveness of these invasive techniques in the improvement of neurophysiological parameters in patients with low back pain with irradiation in the lower extremity, presence of hernias and/or protrusions. Taking into account the good empirical results found in private clinics and the precedents of other studies carried out with short-term follow-up in other regions, this treatment approach of outpatient application in primary care centers could mean a discharge of patients who are referred to the hospital for medical care, imaging tests and surgical interventions.

DETAILED DESCRIPTION:
Low back pain or lumbar pain is the most frequent cause of incapacity for work in Spain, occupying first place among the most common pathologies diagnosed in this country, followed by cervical pain. Non-specific low back pain is the main cause of public spending on health care and labor concepts, with a prevalence of 80%. Furthermore, this pathology represents more than half (52.92%) of the diagnoses of chronic pain that is neither oncologic nor neuropathic. This situation generates high economic, health care and labor costs, representing an equivalent cost of between 1.7% and 2.1% of the Gross Domestic Product.

Low back pain is described as pain located between the lower limit of the ribs and the lower limit of the buttocks, the intensity of which varies according to posture and physical activity, and which is usually accompanied by painful limitation of movement. Approximately 40% of patients with low back pain present irradiation in the lower extremity. The chronification of low back pain can result in central sensitization, causing hypersensitivity to non-painful and painful stimuli even long after the onset of the acute episode of low back pain.

The approach to low back pain offers options such as the administration of drugs, prescription of physical exercise, pain education and modification of patients' habits. Minimally invasive techniques in the management of low back pain are arousing greater interest due to their great advantages. In the field of physical therapy, novel techniques have been developed in recent years, such as ultrasound-guided percutaneous musculoskeletal electrolysis and ultrasound-guided percutaneous neuromodulation, in which different types of electric current are applied through solid needles. Different mechanisms of action have been associated with these invasive techniques, such as a potential effect on the activation of descending pain inhibitory system pathways, the reduction of evoked motor potentials and an increase in intracortical inhibition, suggesting benefits in patients with central sensitization. The invasive techniques of electrolysis and neuromodulation have been applied in other studies at the nervous level, especially in the sciatic nerve at the piriformis and ischiotibial level, in the popliteal fossa and in the foot. It has given good results in lumbar pain. However, there is no study carried out in patients with low back pain and the presence of hernias or protrusions, nor is there any control of the evolution in the medium and long term.

The application of percutaneous neuromodulation has the capacity to modulate neuronal activity in the primary motor cortex, promoting transient and long-term neuroplastic effects. The modulation of this region is related to a decrease in pain due to the relationship with pain processing areas, such as the thalamus, cingulate cortex and periaqueductal gray matter. Electrical stimulation of the peripheral nervous system percutaneously activates a complex neural network that in turn involves a series of neurotransmitters and receptors, such mechanisms being able to promote segmental analgesia and extra-segmental analgesia. Some studies suggest that percutaneous neuromodulation therapy may have a possible beneficial effect in patients with central sensitization, producing improved conditioned pain modulation, reduced motor evoked potential and enhanced intracortical inhibition.

To the authors' knowledge, there are no studies that prove the effectiveness of these invasive techniques in the improvement of neurophysiological parameters in patients with low back pain with irradiation in the lower extremity, presence of hernias and/or protrusions. Taking into account the good empirical results found in private clinics and the precedents of other studies carried out with short-term follow-up in other regions, this treatment approach of outpatient application in primary care centers could mean a discharge of patients who are referred to the hospital for medical care, imaging tests and surgical interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or more than 18 years old.
* Have a medical diagnosis of low back pain with or without radicular involvement and irradiation of symptoms in the lower extremity, by the specialist of the Neurophysiology Service of the Hospital de Terrassa "Consorci Sanitari de Terrassa" or of the Hospital Clínico Universitario de Zaragoza, with confirmation of neurophysiological study, in any of its stages.
* Have access and be able (or have help) to use an online platform to conduct "meetings" with the health professional.
* Read the informed consent and understand the objectives and development of the study.

Exclusion Criteria:

* Be pending compensation or litigation for health problems.
* Receiving physiotherapeutic treatment in the region in the month prior to the study.
* Present severe diseases that may be related to the clinical results: malignancy or history of cancer, tumors or fractures in the region to be treated, blood dyscrasia, severe trauma in the previous 3 months, surgery in the region in the previous 12 months.
* Present contraindications to the therapeutic approach such as: Belonephobia (fear of needles), coagulation alteration, history of adverse reactions, patients reluctant to this type of treatment.
* Subjects who have previously received percutaneous neuromodulation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Present Pain Intensity (NPRS 0-10) | Baseline; 1 month follow-up; 6 month follow-up
  The intensity of hand pain will be recorded, using an 11-point numerical scale (NPRS) (0=no pain, 10=maximum pain). They will be asked for current pain. Because there is no value that determines the minimum clinically relevant difference in hand pain, a 2-point change, or 30% change, will be considered clinically relevant

SECONDARY OUTCOMES:
Change in Neurophysiological study (m/s) | Baseline; 1 month follow-up; 6 month follow-up
  The procedures will be performed by a neurophysiologist with more than 10 years of clinical and research experience using an electroneurogram (needles, electrodes and nerve conduction information processors). The electrophysiological diagnostic criteria for low back pain and lumbar nerve root involvement of the American Association of Neuromuscular and Electrodiagnostic Medicine and the normal ranges of motor and sensory nerve conduction as described in the literature will be used. The following will be taken as study variables: existence of denervation, distal motor latency of the sciatic nerve, distal sensory latency of the sciatic nerve, conduction velocity, action potential amplitude.
Change in straight leg elevation test (range of motion) | Baseline; 1 month follow-up; 6 month follow-up
  The straight leg elevation test will be used to determine the mechanosensitivity of the sciatic nerve. In this test, a structural differentiation of the symptoms will be made at a distance from the area of symptom onset. Performing an internal rotation of the hip if the symptoms are distal (below the knee) or with a dorsiflexion of the ankles if the symptoms are proximal. This test has obtained consistent values in patients with low back pain, with good inter-examiner reliability in its application.
Roland Morris disability Questionnaire | Baseline; 1 month follow-up; 6 month follow-up
  Questionnaire to determine the degree of physical disability derived from low back pain. A self-administered questionnaire consisting of 24 sentences in which the patient has to indicate whether they relate to his or her current situation or not. Score from 0 to 24.
Change in Global rating of change scale | Baseline; 1 month follow-up; 6 month follow-up
  Scale of global change perceived by the patient, designed to detect improvement or deterioration of the patient over time. An 11-point numerical scale (-7=evolving to much worse; +7=fully recovered). Considering +4 and +5 moderate positive changes and +6 and +7 notable changes.
Change in lower extremity strength (Newtons) | Baseline; 1 month follow-up; 6 month follow-up
  The strength of the affected lower extremity will be measured with a hand-held dynamometer (MicroFET 2). The functional movements of hip flexion and extension, knee flexion and extension and ankle flexion and extension will be measured. Three measurements per movement will be taken and the average of them will be obtained.
Change in Sensitivity (discrimination of two points) | Baseline; 1 month follow-up; 6 month follow-up
  The discrimination of two points on the back of the thigh, on the front and back of the leg and the entire region of the foot and ankle will be assessed with a digital caliper. Pressure will be applied with one or two points until causing some discomfort to the patient, having to discriminate whether the patient is stimulated with 1 or 2 points, the minimum distance that he/she manages to discriminate will be recorded. With the patient lying down with eyes closed, the patient will be asked to say "one" when he/she feels that he/she is touched with one point and "two" when he/she feels that he/she is touched with two points.
Change in Sensitivity (Semmes-Weinstein Monofilament Test) | Baseline; 1 month follow-up; 6 month follow-up
  Stimulation by means of pressure filaments, seeking to detect the sensitive threshold by means of 1-second pressures, the necessary pressure will be applied to cause a slight deformation of the filament. The numbers of the filaments (1.65-6.65) of Semmes-Weinstein Monofilament, correspond to a logarithmic function of the equivalent forces (0.0045-447 g). The lightest filament detected will be recorded. With the patient lying down, eyes closed, the subject is asked to verbally signal the moment he/she feels the stimulus in the region to be explored. The filament will be applied vertically over the assessment point, slowly, until the filament bends.
Change in Inhibitory modulation conditioned by pain (Kpa) | Baseline; 1 month follow-up; 6 month follow-up
  It will be performed with the aim of exploring the descending inhibitory pathway. In a first term, the test of pain thresholds by pressure in the affected area is performed. A remote area, usually the arm or hand, is subjected to a painful stimulus (ice cube) or ischemia cuff (maximum 10 min at 200 mmHg or up to VAS 6). At that time, the pressure pain threshold test is repeated on the affected area. An increase in the value of the pressure threshold test will denote a correct functioning of the inhibitory modulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain